CLINICAL TRIAL: NCT03989739
Title: A Cost Effectiveness Analysis of Robotic Versus Laparoscopic Distal Pancreatectomy
Status: Completed | Type: Observational
Sponsor: Fundación de investigación HM (Other)
Responsible Party: Sponsor
Other Study IDs: Fundacionhm
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Surgery
Keywords: Cost-effectiveness; Pancreatectomy; Willingness to pay; Robotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- robotic distal pancreatectomy
  Interventions: Device: Da Vinci
- laparoscopic distal pancreatectomy

INTERVENTIONS:
Device: Da Vinci
  Groups: robotic distal pancreatectomy

SUMMARY:
This is a clinical and cost-effectiveness analysis within a retrospective comparative study of RDP and LDP conducted at Sanchinarro University Hospital from 2011 to 2017. Outcome parameters included surgical and post-operative costs, quality adjusted life years (QALY), and incremental cost per QALY gained or the incremental cost effectiveness ratio (ICER). A sensitivity analysis was carried out in order to propagate the uncertainty of the estimations to the results of the model. The investigators use a multivariate and stochastic sensitivity analysis performed by 5000 Monte Carlo simulations. The cost-effectiveness plane was used to represent all pairs of solutions of the model.

ELIGIBILITY:
Inclusion Criteria:

* Patients (aged over 18 years) with benign or malignant mass without evidence of major vessel involvement were included.
* The indication for resection was given in the context of a multidisciplinary institutional committee

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was carried out at the General Surgery Department of Sanchinarro University Hospital of Madrid.
  Details of the procedure have been described in a previous report and standardized in both groups. RDP was performed using a da Vinci Robotic Surgical System model Si and Xi (Intuitive Surgical, Sunnyvale, CA, USA) (8). All consecutive cases were conducted by the same group of 6 surgeons all with considerable experience in both laparoscopic and robotic approaches.
  Patients (aged over 18 years) with benign or malignant mass without evidence of major vessel involvement were included and assigned either to RDP or LDP, depending on the availability of the robot. The indication for resection was given in the context of a multidisciplinary institutional committee.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Quality-adjusted life years | 2014-2018
  Quality-adjusted life years
ICER | 2014-2018
  Incremental Cost-effectiveness Ratio
Costs | 2014-2018
  Direct costs

IPD SHARING:
Plan to Share IPD: No